CLINICAL TRIAL: NCT04704739
Title: A Phase 1, Open-label Study to Investigate the Pharmacokinetics and Metabolism of GLPG1205 in Healthy Male Subjects Following Single Intravenous [14C]-GLPG1205 Microtracer and Single Oral [14C]-GLPG1205 Administration
Brief Title: Evaluation of Mass Balance and Absolute Bioavailability of GLPG1205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG1205-CL-109; 2020-004550-29 (EudraCT Number)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1205

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG1205 oral and [14C]-GLPG1205 IV (Experimental): Single oral dose of GLPG1205 followed by [14C]-GLPG1205 solution for infusion
  Interventions: Drug: GLPG1205 film-coated tablets; Drug: [14C]-GLPG1205 solution for infusion
- [14C]-GLPG1205 capsule (Experimental): Single oral dose of GLPG1205 as solid formulation
  Interventions: Drug: GLPG1205 capsules

INTERVENTIONS:
Drug: GLPG1205 film-coated tablets — Single oral dose of GLPG1205
  Arms: GLPG1205 oral and [14C]-GLPG1205 IV
Drug: [14C]-GLPG1205 solution for infusion — A 15-minute IV infusion of [14C]-GLPG1205
  Arms: GLPG1205 oral and [14C]-GLPG1205 IV
Drug: GLPG1205 capsules — Single oral dose of GLPG1205 as solid formulation
  Arms: [14C]-GLPG1205 capsule

SUMMARY:
A study in healthy male volunteers to assess how the radiolabelled test medicine is taken up and broken down by the body when given by short infusion into a vein and when given by the mouth in the form of a capsule or tablet.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18-64 years of age (extremes included) (Part 1) and between 45-64 years of age (extremes included) (Part 2), on the date of signing the informed consent form.
* A body mass index (BMI) between 18.0-32.0 kg/m2, inclusive.
* Having a regular (at least) daily defecation pattern (i.e. 1 to 3 times per day).

Exclusion Criteria:

* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. Occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, cannot participate in the study.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability (F) (%) | Between Day 1 and Day 22
  To determine the absolute bioavailability of an oral dose of GLPG1205 relative to an intravenous (i.v.) microtracer dose of [14C]-GLPG1205
Recovery of total radioactivity in urine and feces measured as amount of [14C]-GLPG1205 excreted as percentage of the administered dose (Ae%) | Between Day 1 and Day 22
  To assess the mass balance recovery after a single oral dose of [14C]-GLPG1205

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Tankisheva, MD, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No